CLINICAL TRIAL: NCT01977248
Title: Sensorimotor Affect Relationship-based Therapy (SMART) for Children With Autism Spectrum Disorders Ages 2-12
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Kelly Tanner, Occupational Therapy Research Coordinator, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-00460
Record Dates: First submitted 2013-10-14; First posted 2013-11-06 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Autism Spectrum Disorder; Autistic Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SMART therapy (Experimental): The Sensorimotor Affect Relationship-based Therapy (SMART) program is an interdisciplinary program that teaches children ages 2-12.5 the fundamental skills necessary to build and maintain relationships. Sessions last for 12 weeks at a time and address skills such as: tolerance for sitting and structure, joint attention, eye contact, transitions between activities, participation in group activities, communication skills, and play skills.
  Interventions: Behavioral: Sensorimotor Affect Relationship-based Therapy (SMART)

INTERVENTIONS:
Behavioral: Sensorimotor Affect Relationship-based Therapy (SMART) — The SMART Program is an interdisciplinary program that teaches children ages 2-12.5 the fundamental skills necessary to build and maintain relationships. Sessions last for 12 weeks at a time and address skills such as: tolerance for sitting and structure, joint attention, eye contact, transitions between activities, participation in group activities, communication skills, and play skills.

SUMMARY:
The SMART Program at Nationwide Children's Hospital is an interdisciplinary social skills group that teaches children with autism spectrum disorders (ASD) ages 2-12 the fundamental social skills necessary to build and maintain relationships. The manualized curriculum addresses skills such as joint attention, eye contact, play, and peer engagement. Currently individual goals are set for each child who participates and this is documented in the daily treatment note. In order to research group outcomes, the investigators will use parent questionnaires (an addition to current clinical practices) to measure changes in behavior after each 12 week session for up to one year of treatment. The investigators hypothesize that maladaptive behaviors will decrease and adaptive behaviors will increase in children with ASD after participation in the SMART program.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 to 12.5
* Diagnosis of ASD OR who meet a minimum ASD cutoff score on a screening questionnaire (SCQ or ASQ:SE, depending on age)

Exclusion Criteria:

* Non-English speaking
* Uncorrected vision disorder
* Moderate to severe hearing loss
* Non-ambulatory
* Previous participation in a SMART group
* Accompaniment by aide
* Extreme behavioral disorder

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pervasive Developmental Disorder Behavior Inventory (PDDBI) | Upon enrollment in the study (baseline), day 1 of treatment, and end of treatment for each 12 week session (up to 4 sessions)
  Parent-report questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly J Tanner, MOT, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital Hilliard Close to Home, Hilliard, Ohio, United States